CLINICAL TRIAL: NCT01585142
Title: Assessment of Growth of Infants Fed With BabyNes System (Single-serve Formulas, Adaptative System)
Brief Title: Growth of Infants Fed With BabyNes System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 11.18.INF
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Dietary Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BabyNes system formula (Experimental)
  Interventions: Other: Test formula

INTERVENTIONS:
Other: Test formula — Infant Formulas in powder in single-serve capsules (with a machine for dispensing, four consecutive formulas with customized composition
  Other Names: BabyNes System

SUMMARY:
The purpose of this study is to assess the growth of infants fed with BabyNes System, compared to the World Health Organization Reference, during the first four months of life.

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborn
* Full term newborn (≥ 37 weeks gestation)
* Birth weight ≥ 2500 g and ≤ 4500 g
* Newborn from birth to 14 days of age at the time of enrollment
* The newborn's mother has voluntarily elected to exclusively formula feed her newborn
* Having obtained his/her signed legal representative's informed consentHealthy newborn infant

Exclusion Criteria:

* Congenital illness or malformation that may affect normal growth (especially immunodeficiency)
* Newborn whose mother's BMI was abnormal (<18.5 or >30kg/m2) at start of pregnancy
* Newborn whose mother has diabetes of type-1 or type-2
* Newborn whose mother has a chronic infectious disease
* Newborn whose parents / caregivers cannot be expected to comply with treatment
* Newborn currently participating in another nutritional interventional clinical trial (except for vaccination studies)

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
z-score weight-for-age (WHO Child Growth Standards) | 4 months

SECONDARY OUTCOMES:
Growth | 12 months
  BMI for age z-scores, weight for length z-scores, length for age z-scores, head circumference for age z-scores
Compliance | 12 months
  Volume of formula intake
Morbidity | 12 months
  Number of infants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Spalinger, Dr med., Principal Investigator — Pädiatrische Gastroenterologie und Hepatologie Kinderspital
Locations (4):
- Switzerland (4):
  - Universitäts-Kinderspital beider Basel (UKBB), Basel
  - Hôpital des enfants, Geneva
  - CHUV Unité de Gastroentérologie Pédiatrique DMCP-BH11, Lausanne
  - Pädiatrische Gastroenterologie und Hepatologie Kinderspital, Lucerne